CLINICAL TRIAL: NCT06364137
Title: Engagement and Clinical Impact of the Teleo Virtual Therapy Platform
Brief Title: Engagement and Clinical Impact of the Teleo Virtual Therapy Platform in Clinical Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); MainSquare Co. (dba 'Teleo') (Unknown)
Responsible Party: Principal Investigator, David Hong, Associate Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 73203; R42MH136878 (NIH)
Record Dates: First submitted 2024-04-08; First posted 2024-04-15 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Anxiety Disorders; Mood Disorders
MeSH Terms: conditions — Anxiety Disorders; Mood Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teleo (Experimental): Participants in this group will under therapy for 4 sessions using the Teleo virtual therapy video platform, sessions will be recorded and questionnaires and clinical data will be measured.
  Interventions: Other: Teleo
- Standard videoconferencing (Active Comparator): Participants in this group will under therapy for 4 sessions using standard video platforms (e.g. zoom or other publicly available product), sessions will be recorded and questionnaires and clinical data will be measured.
  Interventions: Other: Standard videoconferencing

INTERVENTIONS:
Other: Teleo — Therapist-led psychotherapy sessions implemented within the Teleo virtual therapy platform.
  Arms: Teleo
Other: Standard videoconferencing — Therapist-led psychotherapy sessions implemented in standard (non-Teleo) video platform
  Arms: Standard videoconferencing

SUMMARY:
The research study will examine engagement in telehealth for children undergoing psychotherapy. Specifically, the pilot trial will examine examine patient engagement in Teleo, a virtual therapy platform specifically designed for psychotherapy with youth, as compared to standard video conferencing.

DETAILED DESCRIPTION:
The research study will examine engagement in telehealth for children undergoing psychotherapy. The study in Phase I entails a pilot randomized trial with a goal to enroll 42 families, examining patient engagement in Teleo, a virtual therapy platform specifically designed for psychotherapy with youth, as compared to standard video conferencing.

Engagement will be assessed using well-established measures - PRIME-O (modified) video coding (session 1), MTT-Y/MTTCG (sessions 1, 4) and attendance data (sessions 1-4). Clinicians in the study will deliver therapy to clients for 4 sessions, providing opportunity to measure temporal sustainment of any engagement differences.

ELIGIBILITY:
Inclusion Criteria:

* Receiving psychotherapy with a licensed professional on the Teleo platform
* Likely have at least 12 sessions remaining.
* Diagnosis of a mental health condition by a licensed clinician

Exclusion Criteria:

* Not under treatment with provider using Teleo platform

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
PRIME-O Video Coding Score | Weeks 1, 2, 3, 4
  Assess therapeutic engagement using modified PRIME-O total score, group scores, and individual item sub-scores. Scores range from 0-40, higher scores indicate 'better' outcome.

SECONDARY OUTCOMES:
My Thoughts about Therapy - Caregiver (MTT-CG) engagement questionnaire scores | Post-intervention (at one month)
  Caregivers will complete modified MTT-CG questionnaire to measure engagement across dimensions of the REACH client engagement framework - Relationship, Expectancy, Attendance, Clarity, and Homework. Scores range from 0-105, higher scores indicate 'better' outcome.
My Thoughts about Therapy - Youth (MTT-Y) engagement questionnaire scores | Post-intervention (at one month)
  Youth will complete questionnaires to measure self-reported engagement across dimensions of the REACH client engagement framework - Relationship, Expectancy, Attendance, Clarity, and Homework. Scores range from 0-105, higher scores indicate 'better' outcome.
Attendance during Psychotherapy Sessions | One month
  Instances and frequency of appointment cancellations, appointment no-shows, and/or discontinuation of therapy will be recorded and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: David S Hong, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-03-31): https://cdn.clinicaltrials.gov/large-docs/37/NCT06364137/ICF_000.pdf